CLINICAL TRIAL: NCT03540537
Title: A Randomized Controlled Trial Comparing Quadratus Lumborum Block and Paravertebral Block for Postoperative Analgesia in Laparoscopic Hepatectomy and Open Hepatectomy
Brief Title: A Trial Comparing Quadratus Lumborum Block (QLB) and Paravertebral Block (PVTB) for Postoperative Analgesia in Hepatectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: NFEC-2017-190
Record Dates: First submitted 2018-04-18; First posted 2018-05-30 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-02

CONDITIONS: Quadratus Lumborum Block; Thoracic Paravertebral Block; Postoperative Analgesia; Hepatectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- PCA for Open Hepatectomy (Other): Patient-controlled intravenous analgesia in Open hepatectomy (PCA solution: 2 μg/kg weight sufentanil and 8.96 mg tropisetron mesylate diluted in 100 ml normal saline；PCA parameters: loading dose: 2 ml, background infusion: 2ml/h, bolus: 0.5ml, lockout-time: 15min; PCA duration: 48 hours from the end of suturing)
  Interventions: Other: Patient-controlled intravenous analgesia
- QLB for Open Hepatectomy (Experimental): Bilateral quadratus lumborum block with 20 ml 0.375% ropivacaine each side(maximum total dose 3 mg/kg) combine Patient-controlled intravenous analgesia (same as PCA for Open hepatectomy Arm)
  Interventions: Other: Patient-controlled intravenous analgesia; Other: Quadratus Lumborum Block
- TPVB for Open hepatectomy (Experimental): T6+T8 of thoracic paravertebral block with 15 ml 0.375% ropivacaine each segment (maximum total dose 3 mg/kg) combine Patient-controlled intravenous analgesia (same as PCA for Open hepatectomy Arm)
  Interventions: Other: Patient-controlled intravenous analgesia; Other: Thoracic Paravertebral Block
- PCA for Laparoscopic Hepatectomy (Other): Patient-controlled intravenous analgesia in Laparoscopic hepatectomy (same as PCA for Open hepatectomy Arm)
  Interventions: Other: Patient-controlled intravenous analgesia
- QLB for Laparoscopic Hepatectomy (Experimental): Bilateral quadratus lumborum block 20 ml 0.375% ropivacaine each side(maximum total dose 3 mg/kg) combine Patient-controlled intravenous analgesia (same as PCA for Open hepatectomy Arm)
  Interventions: Other: Patient-controlled intravenous analgesia; Other: Quadratus Lumborum Block
- TPVB for Laparoscopic Hepatectomy (Experimental): T6+T8 of thoracic paravertebral block with 15 ml 0.375% ropivacaine each segment (maximum total dose 3 mg/kg) combine Patient-controlled intravenous analgesia (same as PCA for Open hepatectomy Arm)
  Interventions: Other: Patient-controlled intravenous analgesia; Other: Thoracic Paravertebral Block

INTERVENTIONS:
Other: Patient-controlled intravenous analgesia — PCIA solution: 2 μg/kg weight sufentanil and 8.96 mg tropisetron mesylate diluted in 100 ml normal saline；PCIA parameters: loading dose: 2 ml, background infusion: 2ml/h, bolus: 0.5ml, lockout-time: 15min; PCA duration: 48 hours from the end of suturing
Other: Quadratus Lumborum Block — Ultrasound-guided Quadratus lumborum block: A broadband (5-8 MHz) convex transducer will be placed transversely in the abdominal flank above the iliac crest to identify the external oblique, internal oblique, transversus abdominis muscles and aponeurosis. Then the external oblique muscle will be followed posteriorly until its posterior border is visualized (hook sign), and the posterior aspect of the Quadratus lumborum muscle is confirmed. A 22-G, 11-mm, short-bevel facet needle will be advanced under direct ultrasound visualization in-plane from anterolateral to postero-medial. Then the 20 ml of 0.375 % ropivacaine will be injected into the lumbar inter-facial triangle (LIFT) behind the quadratus lumborum muscle using hydro-dissection.
  Arms: QLB for Laparoscopic Hepatectomy; QLB for Open Hepatectomy
Other: Thoracic Paravertebral Block — Ultrasound-guided Thoracic paravertebral block: The patient is placed in the lateral position, the spinous processes of T6 and T8 are identified and marks are made 2cm lateral to the spinous processes. The linear(L12-3) probe is placed transversally at the mark to identify the paravertebral space. Then a 22-G needle is inserted in-plane from lateral to medial and advanced until the tip reached the paravertebral space surrounded by the parietal pleura and the superior costotransverse ligament. Then 15 ml 0.375% ropivacaine is injected into the paravertebral space of T6 and T8.
  Arms: TPVB for Laparoscopic Hepatectomy; TPVB for Open hepatectomy

SUMMARY:
Pain after hepatectomy can interfere with the patients' recovery and may contribute to developing long term pain. Opioids, e.g. morphine, fentanyl, sufentanil, works well for postoperative analgesia, but have several side effects such as nausea, vomiting and itching which may be severe enough to affect patients' recovery. In some cases, opioids may cause constipation and urinary retention within the first 24 hours after surgery. Thus, several ultrasound-guided nerve block procedures have been applied to provide postoperative analgesia. Ultrasound-guided thoracic paravertebral block (TPVB) is one of the most used nerve block methods using for post-hepatectomy analgesia. However, in some cases, ultrasound-guided TPVB can cause pneumothorax, hemopneumothorax, and higher block level. The quadratus lumborum block (QLB) is a new developed nerve block which can provide a widespread analgesic effect from T7 to L1. Therefore, this study is to determine whether QLB or TPVB have a better pain control with fewer side effects and complications after laparoscopic and open hepatectomy. The adequate pain control will be assessed by their visual analogue score (VAS) and the postoperative quality of recovery scale (QoR-15, Chinese Version). Additionally, the side effect and complications profile of these two nerve block techniques will also be recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 65 years old for selective hepatectomy from nanfang Hospital, Southern Medical University
* American Society of Anesthesiologists (ASA) risk class I-III;
* Body Mass Index (BMI) is not lesser than 18 and not greater than 30;

Exclusion Criteria:

* Patients refuse to participate
* Allergy to the any agents used in current clinical trial;
* Dependence, tolerance or excessive sensitivity to the anesthetics and psychotropic drugs;
* Patients with nerve block contraindications (e.g. local infection of skin or soft tissue in injection site, serious bleeding tendency or hemorrhagic disease, anatomical aberration which make anesthesiologist cannot perform the ultrasound-guided nerve block, allergic history of local anesthetics, etc.);
* Previous abdominal surgery (except for diagnostic biopsy);
* New York Heart Association (NYHA) classification of cardiac function grade IV and/or Ejection Fraction (EF)≤55%;
* Child-Pugh grading
* Liver function of grade C (Child-Pugh grading)
* Glomerular filtration rate≤60ml/min/1.73m2;
* Obstructive sleep apnea syndrome;
* Chronic obstructive pulmonary disease, asthma, active tuberculosis;
* Cardiac rhythm disorders;
* Past or present history of nervous system diseases and mental disorders (such as epilepsy, Alzheimer's disease, Parkinsonism syndrome, depression,etc.);
* Autoimmune diseases (such as lupus erythematosus, rheumatoid arthritis,etc.)
* Malignant tumors of other systems;
* Other operations are required during the same period;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS | From 1 day before the surgery to the 2 days after surgery
  The visual analogue scale (VAS) is a psychometric response scale which can be used in questionnaires. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points. In current study visual analogue scale is be adopt to assess pain of patients. The VAS ranges from 0-10,0 represents no pain and 10 represents the worst pain.
QoR-15/Quality of Recovery Scale 15(QoR-15) | From 1 day before the surgery to the 2 days after surgery
  The Quality of Recovery-15 scale (QoR-15) is an easy-to-use score for assessing the quality of post-operative recovery. The QoR-15 is a 15-item questionnaire intended to measure QoR after anesthesia and surgery. It comprises five subscales: pain (n = 2), physical comfort (n = 5), physical independence (n = 2), psychological support (n = 2), and emotional state (n = 4) . Each item is scored from 0 to 10, and the possible total score ranges from 0 to 150. A higher total score means better patient QoR.

SECONDARY OUTCOMES:
Total opioids consumption | From admitting in operation room to 48 hours after hepatectomy
  The total amount of opioids consumed during perioperative period
Opioids consumption during hepatectomy Intraoperative opioids consumption | At the end of surgical procedure
  Total doses of opioids consumed during the surgical procedure intraoperatively
Opioids consumption after hepatectomy | Up to 48 postoperative hrs
  Opioids consumption after hepatectomy which are administrated by Patient-controlled intravenous analgesia(PCIA) and by physician's order
First request of analgesia | Up to 48 postoperative hrs
  Time to first request of rescue analgesic drug
Nausea | Up to 48 postoperative hrs
  Incidence of postoperative nausea
Vomiting | Up to 48 postoperative hrs
  Incidence of postoperative vomiting
Respiratory depression | Up to 48 postoperative hrs
  Incidence of postoperative respiratory depression
Pruritus | Up to 48 postoperative hrs
  Incidence of postoperative pruritus
Sedation Score | Up to 48 postoperative hrs
  A score to evaluate patients' sedation deepness Sedation score will be assessed with 'Modified Observer's assessment of alertness/sedation (OAA/S) score'. The OAA/S Scale is composed of the following categories: (1) responsiveness, (2) speech, (3) facial expression, and (4) eyes. The OAA/S Scale can be scored in two ways: the composite score, with a range of 1 (deep sleep) to 5 (alert), in any one of the four assessment categories and the sum of the four component scores, where responsiveness has possible scores of 1, 2, 3, 4 or 5, speech has scores of 2, 3, 4 or 5, and facial expression and eyes have scores of 3, 4 or 5.
Time to first off-bed activity | Up to discharge from hospital
  Postoperative activity
Lower extremity muscle strength | Up to 48 postoperative hrs
  The muscle strength is divided into 6 levels.To observe the flexion of quadriceps.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Tao, MD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Go R, Huang YY, Weyker PD, Webb CA. Truncal blocks for perioperative pain management: a review of the literature and evolving techniques. Pain Manag. 2016 Oct;6(5):455-68. doi: 10.2217/pmt-2015-0012. Epub 2016 May 9. PMID 27156349
- [Background] Wikner M. Unexpected motor weakness following quadratus lumborum block for gynaecological laparoscopy. Anaesthesia. 2017 Feb;72(2):230-232. doi: 10.1111/anae.13754. Epub 2016 Nov 28. PMID 27891579
- [Background] El-Boghdadly K, Elsharkawy H, Short A, Chin KJ. Quadratus Lumborum Block Nomenclature and Anatomical Considerations. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):548-9. doi: 10.1097/AAP.0000000000000411. No abstract available. PMID 27315184
- [Background] Blanco R, Ansari T, Girgis E. Quadratus lumborum block for postoperative pain after caesarean section: A randomised controlled trial. Eur J Anaesthesiol. 2015 Nov;32(11):812-8. doi: 10.1097/EJA.0000000000000299. PMID 26225500
- [Background] Ueshima H, Otake H, Lin JA. Ultrasound-Guided Quadratus Lumborum Block: An Updated Review of Anatomy and Techniques. Biomed Res Int. 2017;2017:2752876. doi: 10.1155/2017/2752876. Epub 2017 Jan 3. PMID 28154824
- [Background] Kadam VR. Ultrasound-guided quadratus lumborum block as a postoperative analgesic technique for laparotomy. J Anaesthesiol Clin Pharmacol. 2013 Oct;29(4):550-2. doi: 10.4103/0970-9185.119148. PMID 24249997
- [Background] Murouchi T, Iwasaki S, Yamakage M. Quadratus Lumborum Block: Analgesic Effects and Chronological Ropivacaine Concentrations After Laparoscopic Surgery. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):146-50. doi: 10.1097/AAP.0000000000000349. PMID 26735154
- [Background] Murouchi T. Quadratus lumborum block intramuscular approach for pediatric surgery. Acta Anaesthesiol Taiwan. 2016 Dec;54(4):135-136. doi: 10.1016/j.aat.2016.10.003. Epub 2016 Dec 9. No abstract available. PMID 27939905
- [Background] Cardoso JM, Sa M, Reis H, Almeida L, Sampaio JC, Pinheiro C, Machado D. [Type II Quadratus Lumborum block for a sub-total gastrectomy in a septic patient]. Braz J Anesthesiol. 2018 Mar-Apr;68(2):186-189. doi: 10.1016/j.bjan.2016.09.009. Epub 2016 Sep 28. PMID 27687315
- [Background] Baidya DK, Maitra S, Arora MK, Agarwal A. Quadratus lumborum block: an effective method of perioperative analgesia in children undergoing pyeloplasty. J Clin Anesth. 2015 Dec;27(8):694-6. doi: 10.1016/j.jclinane.2015.05.006. Epub 2015 Jul 11. No abstract available. PMID 26174113
- [Background] La Colla L, Uskova A, Ben-David B. Single-shot Quadratus Lumborum Block for Postoperative Analgesia After Minimally Invasive Hip Arthroplasty: A New Alternative to Continuous Lumbar Plexus Block? Reg Anesth Pain Med. 2017 Jan/Feb;42(1):125-126. doi: 10.1097/AAP.0000000000000523. No abstract available. PMID 27997495
- [Background] Johnston DF, Sondekoppam RV. Continuous quadratus lumborum block analgesia for total hip arthroplasty revision. J Clin Anesth. 2016 Dec;35:235-237. doi: 10.1016/j.jclinane.2016.08.002. Epub 2016 Sep 26. No abstract available. PMID 27871532
- [Background] Chakraborty A, Khemka R, Datta T. Ultrasound-guided truncal blocks: A new frontier in regional anaesthesia. Indian J Anaesth. 2016 Oct;60(10):703-711. doi: 10.4103/0019-5049.191665. PMID 27761032
- [Background] Visoiu M, Yakovleva N. Continuous postoperative analgesia via quadratus lumborum block - an alternative to transversus abdominis plane block. Paediatr Anaesth. 2013 Oct;23(10):959-61. doi: 10.1111/pan.12240. Epub 2013 Aug 9. PMID 23927552
- [Background] Parras T, Blanco R. Randomised trial comparing the transversus abdominis plane block posterior approach or quadratus lumborum block type I with femoral block for postoperative analgesia in femoral neck fracture, both ultrasound-guided. Rev Esp Anestesiol Reanim. 2016 Mar;63(3):141-8. doi: 10.1016/j.redar.2015.06.012. Epub 2015 Aug 22. English, Spanish. PMID 26302669
- [Background] Lonnqvist PA, Hildingsson U. The caudal boundary of the thoracic paravertebral space. A study in human cadavers. Anaesthesia. 1992 Dec;47(12):1051-2. doi: 10.1111/j.1365-2044.1992.tb04200.x. PMID 1489028
- [Background] Richardson J, Lonnqvist PA, Naja Z. Bilateral thoracic paravertebral block: potential and practice. Br J Anaesth. 2011 Feb;106(2):164-71. doi: 10.1093/bja/aeq378. PMID 21233114
- [Background] Chen H, Liao Z, Fang Y, Niu B, Chen A, Cao F, Mei W, Tian Y. Continuous right thoracic paravertebral block following bolus initiation reduced postoperative pain after right-lobe hepatectomy: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2014 Nov-Dec;39(6):506-12. doi: 10.1097/AAP.0000000000000167. PMID 25304475
- [Background] Pintaric TS, Potocnik I, Hadzic A, Stupnik T, Pintaric M, Novak Jankovic V. Comparison of continuous thoracic epidural with paravertebral block on perioperative analgesia and hemodynamic stability in patients having open lung surgery. Reg Anesth Pain Med. 2011 May-Jun;36(3):256-60. doi: 10.1097/AAP.0b013e3182176f42. PMID 21490523
- [Background] Renes SH, Bruhn J, Gielen MJ, Scheffer GJ, van Geffen GJ. In-plane ultrasound-guided thoracic paravertebral block: a preliminary report of 36 cases with radiologic confirmation of catheter position. Reg Anesth Pain Med. 2010 Mar-Apr;35(2):212-6. doi: 10.1097/aap.0b013e3181c75a8b. PMID 20301827
- [Background] Marhofer P, Kettner SC, Hajbok L, Dubsky P, Fleischmann E. Lateral ultrasound-guided paravertebral blockade: an anatomical-based description of a new technique. Br J Anaesth. 2010 Oct;105(4):526-32. doi: 10.1093/bja/aeq206. Epub 2010 Aug 3. PMID 20685684
- [Background] O Riain SC, Donnell BO, Cuffe T, Harmon DC, Fraher JP, Shorten G. Thoracic paravertebral block using real-time ultrasound guidance. Anesth Analg. 2010 Jan 1;110(1):248-51. doi: 10.1213/ANE.0b013e3181c35906. Epub 2009 Nov 21. PMID 19933536
- [Background] Abdallah FW, Morgan PJ, Cil T, McNaught A, Escallon JM, Semple JL, Wu W, Chan VW. Ultrasound-guided multilevel paravertebral blocks and total intravenous anesthesia improve the quality of recovery after ambulatory breast tumor resection. Anesthesiology. 2014 Mar;120(3):703-13. doi: 10.1097/ALN.0000436117.52143.bc. PMID 24071616
- [Background] Abrahams M, Derby R, Horn JL. Update on Ultrasound for Truncal Blocks: A Review of the Evidence. Reg Anesth Pain Med. 2016 Mar-Apr;41(2):275-88. doi: 10.1097/AAP.0000000000000372. PMID 26866299
- [Background] Pace MM, Sharma B, Anderson-Dam J, Fleischmann K, Warren L, Stefanovich P. Ultrasound-Guided Thoracic Paravertebral Blockade: A Retrospective Study of the Incidence of Complications. Anesth Analg. 2016 Apr;122(4):1186-91. doi: 10.1213/ANE.0000000000001117. PMID 26756911
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Background] Horlocker TT, McGregor DG, Matsushige DK, Schroeder DR, Besse JA. A retrospective review of 4767 consecutive spinal anesthetics: central nervous system complications. Perioperative Outcomes Group. Anesth Analg. 1997 Mar;84(3):578-84. doi: 10.1097/00000539-199703000-00021. PMID 9052305
- [Background] Page A, Rostad B, Staley CA, Levy JH, Park J, Goodman M, Sarmiento JM, Galloway J, Delman KA, Kooby DA. Epidural analgesia in hepatic resection. J Am Coll Surg. 2008 Jun;206(6):1184-92. doi: 10.1016/j.jamcollsurg.2007.12.041. Epub 2008 Apr 14. PMID 18501817
- [Background] Clarke H, Chandy T, Srinivas C, Ladak S, Okubo N, Mitsakakis N, Holtzman S, Grant D, McCluskey SA, Katz J. Epidural analgesia provides better pain management after live liver donation: a retrospective study. Liver Transpl. 2011 Mar;17(3):315-23. doi: 10.1002/lt.22221. PMID 21384514
- [Background] Schreiber KL, Chelly JE, Lang RS, Abuelkasem E, Geller DA, Marsh JW, Tsung A, Sakai T. Epidural Versus Paravertebral Nerve Block for Postoperative Analgesia in Patients Undergoing Open Liver Resection: A Randomized Clinical Trial. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):460-8. doi: 10.1097/AAP.0000000000000422. PMID 27281726
- [Background] Abdelsalam K, Mohamdin OW. Ultrasound-guided rectus sheath and transversus abdominis plane blocks for perioperative analgesia in upper abdominal surgery: A randomized controlled study. Saudi J Anaesth. 2016 Jan-Mar;10(1):25-8. doi: 10.4103/1658-354X.169470. PMID 26955306
- [Background] Blanco R, Ansari T, Riad W, Shetty N. Quadratus Lumborum Block Versus Transversus Abdominis Plane Block for Postoperative Pain After Cesarean Delivery: A Randomized Controlled Trial. Reg Anesth Pain Med. 2016 Nov/Dec;41(6):757-762. doi: 10.1097/AAP.0000000000000495. PMID 27755488